CLINICAL TRIAL: NCT07262567
Title: A Multicenter, Open-Label, Randomized Controlled Phase III Study to Compare the Efficacy and Safety/Tolerability of GFH375 Monotherapy Versus Investigator's Choice of Chemotherapy in Patients With Previously Treated KRAS G12D-Mutant Metastatic Pancreatic Cancer
Brief Title: Phase III Study to Compare GFH375 and Chemotherapy in Patients With KRAS G12D-Mutant Metastatic Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genfleet Therapeutics (Shanghai) Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GFH375X1301
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Fluorouracil; Leucovorin; Tegafur; gimeracil; potassium oxonate; Gemcitabine; Injections; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Experimental group: GFH375; Control group: investigator's choice of Chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GFH375 (Experimental): GFH375, Oral tablets
  Interventions: Drug: GFH375
- Chemotherapy (Active Comparator): There are three chemotherapy regimens. If participants are randomized to the control group, they will receive the treatment as determined by the investigator.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: GFH375 — The experimental group receives GFH375 monotherapy, QD, orally
  Arms: GFH375
Drug: Chemotherapy — The control group includes three treatment regimens: AG, nal-IRI + 5-FU/LV, and S-1. If participants are randomized to the control group, they will receive the treatment which is determined by the investigator.
  Other Names: Irinotecan Hydrochloride Liposome Injection; Fluorouracil Injection; Calcium Folinate; Tegafur,Gimeracil and Oteracil Potassium Capsules; Gemcitabine Hydrochloride for Injection; Paclitaxel for Injection(Albumin Bound)
  Arms: Chemotherapy

SUMMARY:
This study plans to enroll participants with previously treated metastatic pancreatic cancer and harbor centrally confirmed KRAS G12D mutation. These participants are required to experience disease progression on or after at least one prior standard systemic therapy containing fluorouracil or gemcitabine, and either progressed on or were intolerant to the last treatment. Eligible participants will be randomized 1:1 to the experimental group or the control group for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and sign the informed consent form.
* Male or female aged 18-80 years (inclusive) at the time of signing the informed consent form.
* Pathologically confirmed pancreatic cancer (derived from pancreatic ductal epithelium) at metastatic stage.
* Have received at least one prior standard systemic therapy.
* Participants must have at least one measurable lesion (per RECIST 1.1 criteria).
* Expected survival time ≥ 12 weeks as judged by the investigator.
* Have adequate organ function

Exclusion Criteria:

* Other malignant tumors that progressed or required treatment within 3 years prior to randomization.
* With active central nervous system (CNS) metastasis.
* Previous receipt of therapy targeted for KRAS G12D or pan-RAS/KRAS.
* Received radiotherapy within 4 weeks prior to randomization or other local anti-tumor therapy within 4 weeks prior to randomization.
* Received other anti-tumor therapy within 28 days or 5 half-lives (whichever is shorter) prior to randomization.
* With clinically significant severe cardiovascular diseases.
* Stroke or other severe cerebrovascular diseases within 6 months prior to randomization.
* Complicated with major acute or chronic infectious diseases.
* Have severe mental or psychological diseases, or a history of drug abuse or severe alcoholism.
* Pregnant or lactating females.
* Other conditions deemed inappropriate for participation in the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
OS | Up to approximately 2 years
  Overall Survival
PFS | Up to approximately 2 years
  Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1, as Determined by BICR

SECONDARY OUTCOMES:
PFS | Up to approximately 2 years
  Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1, as Determined by investagors
ORR | Up to approximately 2 years
  ORR assessed by investigators and BICR
DCR | Up to approximately 2 years
  DCRassessed by investigators and BICR
DoR | Up to approximately 2 years
  DoR assessed by investigators and BICR
TTR | Up to approximately 2 years
  TTR assessed by investigators and BICR
The incidence and severity of AEs and SAEs | Up to approximately 2 years
  The incidence and severity of AEs and SAEs
EORTC QLQ-C30 Score | Up to approximately 2 years
  Changes in EORTC QLQ-C30
EORTC QLQ-PAN26 Score | Up to approximately 2 years
  Changes in EORTC QLQ-PAN26 Scores
Plasma concentrations of GFH375 | Up to approximately 2 years
  Plasma concentrations of GFH375

IPD SHARING:
Plan to Share IPD: Undecided